CLINICAL TRIAL: NCT03056261
Title: The Effect of Combined General-epidural vs General Anaesthesia on Postoperative Intestinal Function Recovery and Infection in Neonates and Infants Undergoing Gastrointestinal Surgery: a Prospective, Randomised, Controlled Trial
Brief Title: The Effect of Combined General-epidural vs General Anaesthesia on Postoperative Gastrointestinal Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bnai Zion Medical Center (Other Government)
Responsible Party: Principal Investigator, MOSTAFA.SOMRI, Prof Mostafa Somri, Bnai Zion Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BnaiZionMC-16-MS-004
Record Dates: First submitted 2017-02-12; First posted 2017-02-17 (Actual); Last update posted 2017-02-20 (Actual); Status verified 2017-02

CONDITIONS: Epidural Anesthesia; Infection; Infant, Newborn, Diseases
Keywords: Combined general-epidural anesthesia intestinal recovery
MeSH Terms: conditions — Infections; Infant, Newborn, Diseases | interventions — Injections, Epidural; Anesthesia, General

STUDY DESIGN:
Intervention Model Description: comaring combined general anesthesia and epidural technique to general anaesthsia alone or gastrointestinal recovery and pain managment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combined general and epidural (Experimental): Combined general and epidural anesthesia in infants UNDERGOING INTESTINAL SURGERY
  Interventions: Procedure: Combined general and epidural
- General anaesthesia (Placebo Comparator): General anesthesia in infants UNDERGOING INTESTINAL SURGERY
  Interventions: Procedure: General anaesthesia

INTERVENTIONS:
Procedure: Combined general and epidural — Combined general and epidural anaesthesia
  Arms: Combined general and epidural
Procedure: General anaesthesia — General anaesthesia
  Arms: General anaesthesia

SUMMARY:
Sixty neonates and infants will be enrolled and randomised into two groups of n=30 each . For their surgical procedures, one group general (GA) anaesthesia the second group will receive a combined general and epidural anaesthesia (CGEA).

Anaesthetic technique:

Patients in the GA group will be induced with intravenous propofol (2-4 mg.kg-1) and fentanyl (2-4 µg.kg-1) and will receive rocuronium bromide (0.5 mg.kg-1) to facilitate endotracheal intubation. Anaesthesia will be maintained with sevoflurane (2-3%) in an air/oxygen mixture as well as intravenous fentanyl as required.

In the (CGEA) 0.5 ml.kg-1 of 0.25% bupivacaine will be injected into the epidural catheter, followed by a continuous infusion of 0.1% bupivacaine at a rate of 0.2 mg.kg-1.hr-1 for up to 48 hours postoperatively. Assessment of anaesthetic efficacy will be measured Intraoperative care vital signs. And will continuously be monitored with a Datex AS/3 (Engestrom®, Helsinki, Finland) monitor.

The use of antibiotic prophylaxis will be determined by the degree of bowel contamination during surgery, with the commonest regimen consisting of penicillin, gentamicin and metronidazole will be administered. Antibiotics will be continued for 36-48 hours postoperatively to prevent infection arising from the disturbed bowel flora.

Postoperative care, following surgery, will be conducted. The feeding volume will be increased in steps as long as the volume of regurgitated fluid will be less than 20% of the administered breast milk or formula volume. Full feeding will define as oral tolerance of at least 80% of daily maintenance volume. In cases of abdominal distension or vomiting, feeding will withheld until symptom resolution. The nasogastric tube will be removed on bowel function restoration The CRIES score will be use to assess the severity and duration of postoperative pain during the patients' NICU stay. If the CRIES score is ≥4, fentanyl will be continuously intravenously infused in both study group. Fentanyl will be also administered to CGEA patients who experienced pain despite a continuous epidural infusion at 1-5 µg.kg-1.h-1. The amount of fentanyl required for adequate postoperative pain relief will be recorded in both groups.

DETAILED DESCRIPTION:
After approval off the local Ethical Committee of Bnai Zion Hospital, Haifa, Israel and informed parental consent obtained for each participant. Sixty small infants who undergoing GI surgery will be enrolled in this study.

The inclusion criteria are neonates or infants requiring the following major intestinal procedures: duodenoduodenostomy or duodenojejunostomy for duodenal atresia, ileocaecal resection for intestinal volvulus, ileostomy or colostomy closure for congenital anorectal malformations, and corrective surgery for Hirschsprung's disease. The exclusion criteria are concurrent coagulopathies, sepsis, vertebral column malformations, neurological disease, immunocompromise with or without leukopenia, and intestinal necrotising enterocolitis. Patients will be also excluded if they will require exploratory laparotomy or emergent intestinal surgery.

Sixty premature, ex-premature, and full-term neonates and infants meeting the above criteria will enrolled in the study, patients will randomised into two groups of n=30 each ( according to a computer program ) . For their surgical procedures, the first group will receive general anesthesia (GA group), whereas the second group receive combined general and epidural anesthesia (CGEA group).

Anesthetic technique Patients in the GA group will be induced with intravenous propofol (2-4 mg.kg-1) and fentanyl (2-4 µg.kg-1) and receive rocuronium bromide (0.5 mg.kg-1) to facilitate endotracheal intubation. Anaesthesia will be maintained with sevoflurane (2-3%) in an air/oxygen mixture as well as intravenous fentanyl as required.

Patients in the CGEA group will be induce as above in addition to receiving epidural anaesthesia as follows: A 20G epidural catheter (B. Braun Medical Ltd., Melsungen, Germany) through a 19G Crawford epidural needle, so that its tip lays between the desired T5 and T10 spinal segments. Correct catheter placement will be confirmed by portable epidurography after filling the catheter with 0.5 ml iohexol (Omnipaque® 300, Nycomed, Oslo, Norway). A test dose of 0.1 ml.kg-1 of 1% lidocaine with 1:200 000 adrenaline will be administered, and the result and effects on heart rate (HR) and the ST segment will be noted. If the HR increases by at least 20% above baseline and/or ST segment changes will be observed, the catheter will be withdrawl and re positioned. 0.5 ml.kg-1 of 0.25% bupivacaine will be injected into the epidural catheter, followed by a continuous infusion of 0.1% bupivacaine at a rate of 0.2 mg.kg-1.hr-1 for up to 48 hours postoperatively.

Assessment of anesthetic efficacy in both groups will be confirmed by the absence of surges in blood pressure (BP) and HR beyond 20% above baseline. Success of epidural anesthesia will be defined by the correct placement of the epidural catheter between the T5 and T10 spinal segments within two attempts, as well as the obviation for additional systemic analgesia. In cases of epidural technique failure, anesthesia will be maintained by GA and the patient will be removed from the study.

Intraoperative care Intraoperative systolic, diastolic and mean arterial pressures (SBP, DBP, and MAP), HR, arterial oxygen saturation(SaO2), and temperature will be continuously monitored with a Datex AS/3 (Engestrom®, Helsinki, Finland) monitor. All patients in the GA group will mechanically be ventilated, with maintenance of peak inspiratory pressure between 18 and 30 cmH20, and end-tidal CO2 (ETCO2) between 30 and 50 mmHg. Additionally, urine output will be measured at 30-minute intervals.

Two peripheral intravenous cannulae will be inserted preoperatively for each patient, and fluid will be maintained with Ringer's lactate and 5% glucose solutions at 4 ml.kg-1.h-1. Additional Ringer's lactate will be infused for fluid replacement of third-space and/or blood losses. Packed red blood cells will be transfused in cases of blood loss ≥10% of blood volume.

The use of antibiotic prophylaxis will be determined by the degree of bowel contamination during surgery, with the commonest regimen consisting of penicillin, gentamicin and metronidazole will be administered. Antibiotics will continue for 36-48 hours postoperatively to prevent infection arising from the disturbed bowel flora.

Postoperative care following surgery, all patients will be transferred to the neonatal intensive care unit (NICU) where physiological monitoring and mechanical ventilation will continue as appropriate. Blood samples will be collected postoperatively for full blood count, glucose, electrolyte, and blood gas measurement.

The feeding volume will be increased in 5 ml steps as long as the volume of regurgitated fluid is less than 20% of the administered breast milk or formula volume. Full feeding will be defined as oral tolerance of at least 80% of daily maintenance volume. In cases of abdominal distension or vomiting, feeding will withheld until symptom resolution. The nasogastric tube will be removed on bowel function restoration (i.e. defaecation).

The CRIES neonatal postoperative pain score (C=Crying; R=Requires oxygen; I=Increased vital signs; E=Expression; S=Sleepless) [18] will be used to assess the severity and duration of postoperative pain during the patients' NICU stay. Scoring will carried out by the attending nurses every two hours. If the CRIES score is ≥4, fentanyl will be continuously intravenously infused in both study group. Fentanyl will be also administered to CGEA patients who experienced pain despite a continuous epidural infusion at 1-5 µg.kg-1.h-1. The amount of fentanyl required for adequate postoperative pain relief will recorded in both groups.

ELIGIBILITY:
Inclusion Criteria:

* Neonates or infants requiring the following major intestinal procedures: duodenoduodenostomy or duodenojejunostomy for duodenal atresia,
* ileocaecal resection for intestinal volvulus,
* ileostomy or colostomy closure for congenital anorectal malformations,
* corrective surgery for Hirschsprung's disease. emergent intestinal surgery.

Exclusion Criteria:

* The exclusion criteria are concurrent coagulopathies,
* sepsis,
* vertebral column malformations,
* neurological disease,
* immunocompromise with or without leukopenia,
* intestinal necrotising enterocolitis.
* Patients will be also excluded if they required exploratory laparotomy or or emergent intestinal surgery

Ages: 1 Month to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2017-04 (Estimated); Primary Completion 2017-06 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Postoperative intestinal function recovery for neonates and infants undergoing gastrointestinal surgery. Which anesthetic method be superior and favoured as normal practice general or combined general and epidural anesthesia. | upto 20 days postoperative
  The outcomes measured to determine recovery of intestinal function recovery:
  1. Time to first postoperative defecation measured in hours or days
  2. Duration of nasogastric feeding measured in hours or days
  3. Time to tolerance of full oral feeding measured in hours or days

SECONDARY OUTCOMES:
Rate and sort of postoperative infection | upto 20 days postoperative
  1. Surgical site infection (SSI)
  2. Remote site infection (RSI)

CONTACTS AND LOCATIONS:
Overall Officials: Mostafa Somri, M.D., Principal Investigator — Bnai Zion Medical Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gannam-Somri L, Matter I, Hadjittofi C, Vaida S, Khalaily H, Hossein J, Somri M. Combined epidural-general anaesthesia vs general anaesthesia in neonatal gastrointestinal surgery: A randomized controlled trial. Acta Anaesthesiol Scand. 2020 Jan;64(1):34-40. doi: 10.1111/aas.13469. Epub 2019 Oct 7. PMID 31506919